CLINICAL TRIAL: NCT02669056
Title: Brainstem Assesment in a Cohort of Very Preterm Babies (Less Than 28 Weeks)
Brief Title: Brainstem and Prematurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-35; RCAPHM15_0265 (Other: APHM)
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Very Premature Infants
MeSH Terms: interventions — Videotape Recording; Growth Charts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- preterm babies (Experimental): preterm babies (less than 28 weeks)
  Interventions: Other: 5-HT measurement; Other: cerebral MRI; Other: Video recording; Other: EEG; Other: growth curves; Other: ASQ questionnaire
- term babies (Other): term babies with blood test prescription
  Interventions: Other: 5-HT measurement

INTERVENTIONS:
Other: 5-HT measurement
Other: cerebral MRI
  Arms: preterm babies
Other: Video recording
  Arms: preterm babies
Other: EEG
  Arms: preterm babies
Other: growth curves
  Arms: preterm babies
Other: ASQ questionnaire
  Arms: preterm babies

SUMMARY:
Although significant advances in neonatal care have increased survival rates of preterm infants born before 28 weeks gestation, a concomitant decrease in neuro developmental disorders has not been achieved. Cerebral injuries, well documented during the previous years, in preterm babies are particularly deleterious since they occur in a developing brain. They affect both white and grey matter by complex mechanisms and the principal targets are the developing oligodendrocytes and neurons of the subplate. All these criteria define the encephalopathy of prematurity. Nevertheless, the consequences of prematurity at the level of the brainstem are not very well known and may explain neuro-developmental disorders with normal MRI.

The assessment of the motor repertoire is complementary to the neurological examination and may represent a diagnostic tool for cerebral palsy, mild motor deficits and delayed acquisition in children. The newborn have a rich motor repertoire. GMs play a key role in the development due to the feedback that they send to cortical neurons and reflect the maturational stage of the Central Nervous System (CNS). Lesions of the brainstem caused by prematurity may induce alterations of the motor repertoire.

Dysautonomic disorders, such as bradycardia, apneas, feeding problems, that occur frequently in very preterm babies reflect brainstem abnormalities. These symptoms are also described in other pathologies, in Rett syndrome and sudden infant death syndrome (SIDS). In these pathologies deficits of the 5-HT system have been described and associated with dysautonomia. It would then be interesting to evaluate 5-hydroxytryptamine (5-HT) levels in very preterm babies.

The serotonergic system develops very early during gestation and is one of the first neurotransmitter to appear in the developing brain. The main 5-HT nuclei are located within the brainstem. 5-HT plays an important role in the homeostasis and the modulation of the respiratory network. Moreover, previous studies have shown that 5-HT projections to the spinal cord are involved in posture and in the coordination. It is tempting to think that 5-HT deficits may have some repercussions on the development of the CNS, changing activity dependent processes, such as spontaneous activity recorded at the spinal level in rodents.

In this project, the 5-HT platelet levels in preterm infants born before 28 weeks will be compared with newborns. a correlation between the levels of 5-HT with MRI of the posterior fossa, GMs and dysautonomia different parameters such as heart rate variability, suction-swallowing and different breathing techniques will be established

ELIGIBILITY:
Inclusion Criteria:

* Birth less than 28 weeks
* known gestational age
* Birth in born
* Infant without genetic syndrom, evolutive neurologic disease, chronic disorder, malformative pathology
* Infant without intra-ventricular haemorrhage with dilatation or intraparenchymal haemorrhage
* Infants without mechanical ventilation

Exclusion Criteria:

• Infant with congenital cardiopathy, congenital brainstem disorder, Pierre Robin sequence

Max Age: 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
5-HT levels | term age (37 weeks)
  5-HT platelets levels will be measured in very preterm and in term infants and compared (5-HT platelets level reflect the central 5HT level.

SECONDARY OUTCOMES:
Posterior fossa injury | at term age (37 weeks)
  MRI will be performed at term age to analyse preterm cerebral structure focusing on the posterior fossa
General movements (GMs) assesment | 3 times in the hospitalization period and at 3 month post-term age
  GMs will be video taped at during the writing movements period and fidgety period and analyzed to detect abnormal GMs
R-R variability assesment | at 36 weeks
  The autonomic nervous system activity level will be assessed by R-R variability analyze during polysomnographic recordings
Respiratory pattern assessment | at 36 weeks
  Respiratory pattern assessment will be analyzed during polysomnographic recordings to detect apneas, sighs…
Ages and Stages Questionnaires (ASQ) | 12 and 24 month post-term age
  ASQ questionnaire as neurodevelopmental assessment will be send to parents
weight and statural growth assessment | until 24 month postterm age
statural growth assessment | until 24 month postterm age
Hospitalization duration | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — APHM
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France